CLINICAL TRIAL: NCT01196702
Title: Investigation of the Lymphocyte Surface Expression of Patients With Primary Immunodeficiency (Common Variable Immunodeficiency (CVID)), Compared to Controls
Brief Title: Lymphocyte Immunophenotyping in Common Variable Immunodeficiency
Status: Completed | Type: Observational
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Principal Investigator, Mathew Buckland, Consultant Immunologist, Barts & The London NHS Trust
Other Study IDs: 006749
Record Dates: First submitted 2010-09-06; First posted 2010-09-08 (Estimated); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Common Variable Immunodeficiency; Granulomatous Disease; Bronchiectasis; Immunoglobulin Treatment
Keywords: common variable immunodeficiency; granulomatous disease; crohns disease; bronchiectasis; immunoglobulin replacement or treatment; B-cell immunophenotyping
MeSH Terms: conditions — Common Variable Immunodeficiency; Bronchiectasis; Crohn Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood serum samples kept for one year in secure laboratory.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- CVID: Patients with common variable immunodeficiency
- CVID and granulomatous disease: Patients with CVID complicated with granulomatous inflammation
- CVID and bronchiectasis: Patients with CVID complicated by bronchiectasis
- Control on Immunoglobulin: Patients on immunoglobulin long-term who do not have an immunodeficiency
- Control bronchiectasis: Controls with bronchiectasis not caused by a known immunodeficiency
- Control with granulomatous disease: Control patients with Crohn's Disease as this is a disease that causes granulomatous inflammation.
- Healthy Controls

SUMMARY:
The purpose of this study is to discover if differences in the surface markers of B-cells (antibody producing cells of the immune system) in Common Variable Immune Deficiency (CVID) are related to CVID or its complications/treatment (e.g. bronchiectasis, granulomatous disease, immunoglobulin treatment).

The study hypothesis is that the altered B-cell surface markers are related to CVID, and not to the complications or treatment of CVID.

DETAILED DESCRIPTION:
Common Variable Immune Deficiency (CVID) is a syndrome containing a spectrum of disorders which results in weakened immunity and recurrent infections. The ESID (European Society for Immunodeficiencies) CVID definition includes patients with marked decrease of IgG (at least 2 standard deviations below the mean for age). Patients must also have disease onset at an age over 2 years, absent isohaemagglutinins and/or response to vaccines and other defined causes of hypogammaglobulinaemia must be excluded. The Euroclass system of classifying CVID is the result of a European multicentre trial attempting to develop a consensus of two existing classification schemes of B-cell immunophenotyping. In this paper it was shown that B-cell immunophenotype correlated with coincidence of clinical sequelae and it suggested implementing this to further classify CVID to give prognostic and therapeutic information. However, it has not yet been shown that these alterations in B-cell immunophenotype are the result of CVID itself and not caused by the treatment or complications of CVID (e.g. immunoglobulin replacement therapy, granulomatous disease, bronchiectasis). The aim of this study is to show that alterations in B-cell immunophenotype are caused by CVID itself and not by its complications or treatment. The study will therefore compare CVID patients to suitable control patients with granulomatous disease, bronchiectasis and on long-term immunoglobulin therapy. A control group of normal people will also be included to ensure the assay can detect normality and to show differences between normal people and patients with CVID.

ELIGIBILITY:
Inclusion Criteria:

* 18 or over
* Competent to consent
* Have diagnosis of Common Variable Immunodeficiency, granulomatous disease, on long term immunoglobulin or bronchiectasis.

Exclusion Criteria:

* Under 18
* Unable to consent.
* Medical problem that could alter B-cell immunophenotype (except for the diagnoses in the inclusion criteria)/

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients selected from medical clinics in the order of attendance with common variable immunodeficiency, bronchiectasis, on long-term immunoglobulin treament and granulomatous disease. Must be able to give consent for testing of B-cell immunophenotype. Healthy control samples taken from colleagues.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Percentage of B-cells of all lymphocytes | 5 months
  Look at percentage of cells within the lymphocyte gate that express the B-cell marker CD19, and compare to healthy controls and non-healthy controls.
Percentage of class switched memory B-cells as a percentage of B-cells | 5 months
  Percentage of class-switched memory B-cells (expressing CD27 and CD19), that do not express IgM or IgD, as a percentage of B-cells. This is reduced in CVID and this will be compared between controls and the patients with CVID.

SECONDARY OUTCOMES:
Percentage expression of CD21 and CD38 | 5 months
  Look for abnormalities in the CVID group and compare to control groups in the numeber of B-cells expressing low levels of CD21 (CD21 lo), and high CD38.

CONTACTS AND LOCATIONS:
Locations (1):
- Barts and the London NHS Trust, London, United Kingdom

REFERENCES:
- [Background] Wehr C, Kivioja T, Schmitt C, Ferry B, Witte T, Eren E, Vlkova M, Hernandez M, Detkova D, Bos PR, Poerksen G, von Bernuth H, Baumann U, Goldacker S, Gutenberger S, Schlesier M, Bergeron-van der Cruyssen F, Le Garff M, Debre P, Jacobs R, Jones J, Bateman E, Litzman J, van Hagen PM, Plebani A, Schmidt RE, Thon V, Quinti I, Espanol T, Webster AD, Chapel H, Vihinen M, Oksenhendler E, Peter HH, Warnatz K. The EUROclass trial: defining subgroups in common variable immunodeficiency. Blood. 2008 Jan 1;111(1):77-85. doi: 10.1182/blood-2007-06-091744. Epub 2007 Sep 26. PMID 17898316